CLINICAL TRIAL: NCT04056650
Title: Data Driven Health Decisions in the Wild: A Platform for Actionable N-of-1 Studies
Brief Title: Assessing the Effectiveness of an N-of-1 Platform Using Study of Cognitive Enhancers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jason Bobe, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: GCO 18-0756
Record Dates: First submitted 2019-08-09; First posted 2019-08-14 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Cognitive Performance
Keywords: N-of-1; Caffeine; L-theanine; Nootropic; Cognition; Individualized
MeSH Terms: interventions — theanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single caffeinated beverage/supplement (Active Comparator)
  Interventions: Dietary Supplement: Caffeine supplement; Device: N1 app
- Combination caffeine and L-theanine (Active Comparator)
  Interventions: Drug: L-theanine; Dietary Supplement: Caffeine supplement; Device: N1 app

INTERVENTIONS:
Drug: L-theanine — up to 250 mg
  Arms: Combination caffeine and L-theanine
Dietary Supplement: Caffeine supplement — 50-400mg
Device: N1 app — N1 App on mobile device

SUMMARY:
The growing consumer-grade molecular and digital wellness market is generating unprecedented volumes of information to support decision-making around individual health. Current trends suggest the demand for personalized health information, tools, and services will continue to rise in the next decade. What is missing is a reliable, individualized way to turn this data into action. Dialogue around consumer health often ignores the disconnect between measurements and goals. For example, monitoring one's weight is not the same as losing weight, and counting steps is not the same as lowering blood pressure. If individuals are to benefit from data, they must be able to relate changes in their personal data to targeted changes in actions and outcomes. There is a great need and opportunity to adapt the tools and capabilities of modern computer science, statistics, and clinical trial design to the needs of individual patients and consumers. The team at the Institute for Next Generation Healthcare (INGH) has created a smartphone-based app ("N1 app") and study platform that together allow individuals to design, implement, and analyze methodologically sound, statistically robust studies of their personal health data. The focus of the platform will be the creation of single-participant randomized crossover studies, known as n-of-1 trials. The platform employs informatics-based intelligence that automates study design and analysis while simultaneously maintaining high standards of statistical rigor and reproducibility.

These novel methods and tools are designed to empower individuals to make rational, data-driven choices about their own health, maximizing the benefit all will receive from new and existing sources of personal health data.

DETAILED DESCRIPTION:
The growing burden of chronic disease in the U.S. and the economics of accountable care are driving a shift toward proactive approaches to disease prevention and health maintenance. At the same time, precision medicine studies continue to reveal substantial heterogeneity in the manifestations of even the most common chronic diseases. The bulk of morbidity and mortality in the U.S. arises from conditions with a significant lifestyle component (e.g. type II diabetes), and responsibility for monitoring and maintaining health largely falls on individuals.

Recent advances in molecular biology, sensors, and digital health technology underlie rapidly growing market availability of products and devices for measuring and monitoring individual health. A vast array of wearable devices, smart home monitors, and health tracking apps provide an unprecedented view of individuals "in the wild" and provide customers with health information once accessible only to researchers. The growing digital health market is generating unprecedented volumes of information to support decision making around individual health, and current trends suggest the demand for personalized health information, tools, and services will continue to grow in the next decade.

What is missing from this technological and scientific growth is a reliable, individualized way to translate data into action. If society wants to prevent diabetes, heart disease, and other chronic illnesses that kill millions of Americans each year, individuals must be empowered to address precursor conditions like obesity, hypertension, and depression. Dialogue around consumer health often fails to address the profound disconnect between measurements and outcomes/goals; e.g. monitoring one's weight is not the same as losing weight, and counting steps is not the same as lowering blood pressure. Data are only useful if they can help individuals identify interventions that work for them. The combination of diet, exercise, drugs/supplements, activities, and lifestyle changes that targets an individual's particular set of health problems is unique to him or her, and it is dependent on a complex web of factors including genetics, environment, and personal lifestyle. If individuals are to benefit from data, they must be able to relate changes in their personal data to targeted adjustments in actions and outcomes. This effectively necessitates conducting a robust trial at the level of the individual to determine the most promising recipe of personal lifestyle adjustments to effect change.

To address these challenges, the researchers have developed a unified statistical framework for producing consistent, interpretable study results from diverse n-of-1 study designs. The analysis framework is the backbone of the initial software platform, which includes modules for study design, e-consent, data ingestion, data analysis, and visualization of results.

To test this platform, the researchers plan to deploy a prototype study that allows individuals to test the cognitive effects of two commonly consumed substances: caffeine and caffeine in combination with a safe, prevalent compound, L-theanine. Each enrolled individual will participate in his/her own n-of-1 trial. After a baseline period where neither treatment is taken, participants will alternate between the two treatments ("caffeine alone" and "caffeine + L-theanine") according to a predefined schedule. Participants will complete a daily cognitive assessment composed of 3 validated cognitive tests administered via the N1 app. The platform will analyze the cognitive assessment data and determine whether there is a statistically meaningful treatment effect for either treatment compared to baseline for any of the 3 cognitive tests for each individual that completes the study.

It is important to state explicitly that the research objectives for this protocol are not related to the efficacy of L-theanine and caffeine. This specific study is designed to allow the researchers to efficiently recruit and enroll subjects so that the underlying statistical methods and software platform for executing n-of-1 trials may be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* US resident
* 18 years old or over
* Has an iPhone
* Regular caffeine drinker

Exclusion Criteria:

* Pregnant/breastfeeding
* Any contraindication/health issue in which risk is added by consumption of caffeine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Percent of individuals who reach study completion | Up to 27 days
  Percent of individuals that complete their n-of-1 trial after study initiation

SECONDARY OUTCOMES:
Percent of completed n-of-1 trials that yield statistically meaningful results. | Up to 27 days
  Percent of individual n-of-1 studies that yield statistically conclusive results, for the comparisons (a) caffeine vs. baseline, (b) L-theanine + caffeine vs. baseline.
Study adherence. | Up to 27 days
  Percent of total actions required for the study (e.g. taking assigned treatments and completing daily cognitive assessment) completed by individual and in aggregate.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Bobe, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bobe JR, Buros J, Golden E, Johnson M, Jones M, Percha B, Viglizzo R, Zimmerman N. Factors Associated With Trial Completion and Adherence in App-Based N-of-1 Trials: Protocol for a Randomized Trial Evaluating Study Duration, Notification Level, and Meaningful Engagement in the Brain Boost Study. JMIR Res Protoc. 2020 Jan 8;9(1):e16362. doi: 10.2196/16362. PMID 31913135